CLINICAL TRIAL: NCT04497376
Title: Prospective Randomized Comparison Between Upgraded '2C3L' vs. PVI Approach for Catheter Ablation of Persistent Atrial Fibrillation
Brief Title: Comparison Between Upgraded '2C3L' vs. PVI Approach for Catheter Ablation of Persistent Atrial Fibrillation
Acronym: PROMPT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Heart Health Research Centre (Unknown); The George Institute for Global Health, China (Other); The George Institute for Global Health, Australia (Other); Fukuoka University (Other)
Responsible Party: Principal Investigator, Chang sheng Ma, Director of Cardiology, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017YFC0908803
Record Dates: First submitted 2020-07-08; First posted 2020-08-04 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Persistent Atrial Fibrillation; Catheter Ablation
Keywords: Pulmonary vein antral isolation; Upgraded '2C3L'; Arrhythmia-free survival
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upgraded '2C3L' (Experimental): Patients randomized to the upgraded '2C3L' arm will first undergo ethanol infusion in the vein of Marshall (EI-VOM) followed by the '2C3L' ablation step which includes bilateral circumferential PV antral ablation and linear ablations across the left atrial roof, mitral isthmus (MI), and cavotricuspid isthmus (CTI).
  Interventions: Procedure: upgraded '2C3L'
- Pulmonary vein antral isolation (PVI) (Active Comparator): Patients randomized to the PVI arm will undergo right PV antrum ablation, followed by the left PVA ablation. Radiofrequency should be applied 1 cm proximal to the PV ostia in a wide-area circumferential pattern. Complete PVI will be achieved when all PV potentials within each antrum recorded by the high-density mapping catheter are abolished.
  Interventions: Procedure: pulmonary vein antral isolation

INTERVENTIONS:
Procedure: upgraded '2C3L' — Patients randomized to the upgraded '2C3L' arm will first undergo EI-VOM, followed by the '2C3L' ablation step. The details include: (1). EI-VOM procedure: An 8.5-French-long sheath or a steerable long sheath is sent to the coronary sinus (CS) via the femoral vein. A JR4.0 catheter is inserted into the CS to identify the ostium of the VOM. Subsequently, a BMW wire supported by an OTW balloon catheter is advanced into the VOM. The balloon is inflated with 6 to 8 atm in the VOM. A selective venogram of the VOM is obtained by slowly injecting 1 mL of contrast medium. Then, ethanol is slowly injected into the VOM and selective venography of the VOM is repeated. (2) . After EI-VOM, radiofrequency ablation was performed to achieve bilateral pulmonary vein isolation and bidirectional block of mitral isthmus line, roof line, and cavotricuspid isthmus line. (3). Any organized AT observed during the procedure will be targeted as well.
  Other Names: EI-VOM+2C3L
  Arms: Upgraded '2C3L'
Procedure: pulmonary vein antral isolation — After reconstructing the left atrial geometry, PVI will be performed (the right PV antrum (PVA) will be ablated first, followed by the left PVA. ) in a wide area circumferential pattern. Complete PVI will be achieved when all PV potentials within each antrum recorded by the high-density mapping catheter are abolished. The endpoint of the circumferential PVA ablation procedure is to achieve electrical bilateral PV isolation, that is, the PV potentials associated with atrial electrical activity cannot be recorded during sinus rhythm or CS pacing (entrance block). A waiting period of at least 20 min (after the last PV is isolated) will be used during which spontaneous PV reconnection will be related. , and tDemonstration of exit block (he by pacing in the PV cannot be and proving the absence of transmitted conduction to capture the atrium) may be performed but is not mandatory. Any organized AT observed during the procedure will be targeted as well.
  Other Names: PVI
  Arms: Pulmonary vein antral isolation (PVI)

SUMMARY:
Catheter ablation has emerged as an important treatment option for patients with symptomatic atrial fibrillation (AF). Pulmonary vein antral isolation (PVI) is now considered the cornerstone technique of AF ablation and has shown promise in treating paroxysmal atrial fibrillation (PAF). However, there is no unique strategy for ablation of persistent AF (PeAF), whether PVI alone is sufficient to prevent patients from recurrence remains controversial. The PROMPT-AF study is a prospective, multicenter, randomized trial involving a blinded assessment of outcomes, which is designed to compare arrhythmia-free survival between PVI and an ablation strategy termed upgraded '2C3L' for ablation of PeAF.

DETAILED DESCRIPTION:
The PROMPT-AF study will include 498 patients undergoing their first catheter ablation of PeAF. All patients will be randomized to either the upgraded '2C3L' arm or PVI arm in a 1:1 fashion. The upgraded '2C3L' technique is a fixed ablation approach consisting of EI-VOM, bilateral circumferential PVI, and three linear ablation lesion sets across the mitral isthmus, left atrial roof, and cavotricuspid isthmus. The follow-up duration is 12 months. The primary endpoint is the rate of documented atrial tachycardia arrhythmias of >30 seconds, without any antiarrhythmic drugs, in 12 months after the index ablation procedure (excluding a blanking period of 3 months).

ELIGIBILITY:
Inclusion criteria

Patients must meet all the following criteria to be included in the study:

1. age between 18 and 80,
2. patients undergoing a first-time ablation procedure for non-valvular AF,
3. patients with defined as a sustained episode more than 3 months
4. PeAF documented by ECG, Holter, loop recorder, telemetry, trans-telephonic monitor or implanted device within 90 days6 months of the ablation procedure,
5. patients experienced symptoms caused by AF and these symptoms include but are not limited to palpitations, presyncope, syncope, fatigue, and shortness of breath,
6. AF refractory to at least one AAD,
7. willingness, ability and commitment to provide informed consent and participate in follow-up evaluations.

Exclusion criteria Patients are to be excluded if any of the following criteria is met：

1. patients with paroxysmal AF,
2. patients with AF secondary to an obvious reversible cause,
3. patients with left atrial diameter ≥ 60 mm in the parasternal long axis view,
4. left ventricular ejection fraction (LVEF) < 30%,
5. patients with triple (aspirin, clopidogrel and OAC) or dual (clopidogrel and OAC) antithrombotic therapy which predispose patients to higher risk of periprocedural bleeding. (e.g., Coronary percutaneous transluminal coronary angioplasty (PTCA)/stenting within the previous 90 days),
6. patients with contraindication to anticoagulation,
7. patients with contraindication to right or left sided heart catheterization,
8. pregnancy,
9. life expectancy less than 1 year (advanced malignant tumor, end stage renal disease, etc.),
10. patients cannot be removed from antiarrhythmic drugs for reasons other than AF.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
The recurrence rate of atrial tachycardia arrhythmias | 1 year
  freedom from any documented atrial arrhythmia after a 3-months post-ablation blanking period, including AF, AT, and AFL, for more than 30 seconds in the absence of antiarrhythmic drug (AAD) therapy.

SECONDARY OUTCOMES:
Freedom from AF/AT with or without AADs | 1 year
  Time to the first occurrence of AF, AT in the presence of AAD therapy after one ablation procedure.
Freedom from AF/AT off AADs | 1 year
  Recurrent AT/AFL over 30 seconds after a 3-month post-ablation blanking period in the absence of AAD
Freedom from AF off AADs | 1 year
  Recurrent AF over 30 seconds after a 3-month post-ablation blanking period in the absence of AAD
AF burden | 1 year
  AF burden (% time) on continuous monitoring during 12 months after the 3-months blanking period,
Freedom from AF/AT after multiple procedures | 1 year
  freedom from any documented atrial arrhythmia (AF, AT, and AFL) of more than 30 seconds, after repeated ablation1 or 2 ablation procedures, including AF, AT, and AFL, for more than 30 seconds on/off AADs.
Incidence of procedural complications | Within 1 month after the procedure
  cardiac tamponade or perforation, phrenic nerve injury, acute coronary occlusion, leading to death, intervention required, or prolonged hospitalization, strokes /thromboembolism related to AF ablation, pulmonary vein stenosis, left atrial oesophageal fistula, and vascular complications requiring intervention (e.g., pseudoaneurysm, arteriovenous fistula).
AFEQT score change between baseline and 12 month | 1 year
  Quality of life assessed by AF effect on quality-of-life (AFEQT) questionaire
EQ5D score change between baseline and 12 month | 1 year
  Quality of life assessed by EuroQol 5-dimension (EQ5D) scale

CONTACTS AND LOCATIONS:
Overall Officials: Caihua Sang, MD, Principal Investigator — Beijing Anzhen Hospital; Changsheng Ma, MD, Principal Investigator — Beijing Anzhen Hospital; Jianzeng Dong, MD, Principal Investigator — Beijing Anzhen Hospital; The First Affiliated Hospital of Zhengzhou University; Chenyang Jiang, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (12):
- China (12):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Taizhou Hospital of Zhejiang Province, Taizhou, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Jiangsu Provincial Hospital, Nanjing, Jiangsu
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Renji Hospital, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Sang C, Liu Q, Lai Y, Xia S, Jiang R, Li S, Guo Q, Li Q, Gao M, Guo X, Huang L, Liu N, Jiang C, Zuo S, Liu X, Li M, Ge W, Song S, Chen L, Xie S, Zou J, Chen K, Liu X, Hu H, Wang X, Zhang J, Wang Z, Wang C, He L, Jiang C, Tang R, Zhou N, Wang Y, Long D, Du X, Jiang C, Macle L, Dong J, Ma C; PROMPT-AF investigators. Pulmonary Vein Isolation With Optimized Linear Ablation vs Pulmonary Vein Isolation Alone for Persistent AF: The PROMPT-AF Randomized Clinical Trial. JAMA. 2025 Feb 4;333(5):381-389. doi: 10.1001/jama.2024.24438. PMID 39556379